CLINICAL TRIAL: NCT05870683
Title: Comparison of the Efficacy of Tegoprazan-containing Versus Esomeprazole-containing Dual Therapy for Helicobacter Pylori Eradication: a Prospective, Multicenter, Randomized Controlled Study （SHARE2301）
Brief Title: Comparison of Two Dual Therapies in the First-line Treatment of Helicobacter Pylori Infection （SHARE2301）
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanqing Li (Other)
Collaborators: Linyi People's Hospital (Other); Weifang Medical University (Other); Zhengzhou Central Hospital (Other); Yuncheng Traditional Chinese Medicine Hospital (Other); The Affiliated Hospital of Qingdao University (Other); The People's Hospital of Jimo (Unknown); Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Vice-President, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHARE2301
Record Dates: First submitted 2023-05-07; First posted 2023-05-23 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — tegoprazan; Amoxicillin; Esomeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 14-day Tegoprazan-Amoxicillin dual therapy (Experimental): 14-day Tegoprazan-Amoxicillin dual therapy, Tegoprazan（Luo Xin Pharmaceutical Group Co. LTD）50mg bid, Amoxicillin (Amoxicillin, United Laboratories Co. LTD) 750mg qid
  Interventions: Drug: Tegoprazan; Drug: Amoxicillin
- 14-day Esomeprazole-Amoxicillin dual therapy (Active Comparator): 14-day Esomeprazole-Amoxicillin dual therapy, Esomeprazole（Astrazeneca Pharmaceutical Co., LTD.) 20mg qid, Amoxicillin (Amoxicillin, United Laboratories Co. LTD) 750mg qid
  Interventions: Drug: Amoxicillin; Drug: Esomeprazole

INTERVENTIONS:
Drug: Tegoprazan — Included in dual eradication medication.
  Arms: 14-day Tegoprazan-Amoxicillin dual therapy
Drug: Amoxicillin — Included in dual eradication medication.
Drug: Esomeprazole — Included in dual eradication medication.
  Arms: 14-day Esomeprazole-Amoxicillin dual therapy

SUMMARY:
Helicobacter pylori (H. pylori) infection is a common global infectious disease of the gastrointestinal tract. Helicobacter pylori eradication can effectively prevent the development of stomach cancer. Progressive application of dual therapy for the eradication of Helicobacter pylori. Tegoprazan, a Potassium-Competitive Acid Blockers. The efficacy of P-CAB agents represented by vonoprazan in H. pylori eradication therapy has been widely verified.

DETAILED DESCRIPTION:
In 1989, it was suggested that amoxicillin combined with PPI could eradicate Hp infection, and in 2015, a prospective, multicenter, randomized controlled study in Taiwan with a large sample showed that the eradication rate of Hp could reach 96.6% with dual therapy for primary treatment of Hp infection, and the results of intention-to-treat analysis were as high as 95.3%. 95.3%. In 2020, a meta-analysis showed that high-dose dual therapy had the same efficacy and fewer side effects than other recommended regimens in first-line treatment. In terms of dosing days, multiple randomized controlled studies and meta-analyses from 2020-2021 have shown that 14 days of high-dose dual therapy is more effective in eradicating H. pylori.

Tegoprazan, a Potassium-Competitive Acid Blockers (P-CAB), is a new type of acid-suppressing drug that compensates for the short half-life of acid-activated traditional acid-suppressing PPI and the low mucosal healing rate due to insufficient acid suppression. The efficacy of P-CAB agents represented by vonoprazan in H. pylori eradication therapy has been widely verified. 2022, tegoprazan was approved by the State Drug Administration for the new indication of eradication of H. pylori infection in adults in combination with appropriate antimicrobial therapy, and its efficacy in clinical application has not yet been verified.

ELIGIBILITY:
Inclusion Criteria:

* Helicobacter pylori infection (either positive for histopathological test, rapid urease test, or C13/C14 urea breath test).
* Patients who have not previously received helicobacter pylori eradication therapy.

Exclusion Criteria:

* Serious underlying diseases, such as liver insufficiency, renal insufficiency, immunosuppression, malignant tumor, coronary heart disease (angina pectoris or coronary artery stenosis ≥ 75%).
* Those who are not willing to take contraceptive measures during pregnancy, lactation or the trial.
* Active gastrointestinal bleeding.
* History of drug allergy.
* History of upper gastrointestinal surgery.
* Medication history of bismuth, antibiotics and PPI within 4 weeks.
* Other behaviors that may increase the risk, such as alcohol and drug abuse.
* Unable or unwilling to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | Immediately after follow-up check
  Both intention to treat (ITT) and per-protocol (PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infections in two groups. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 80% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
Rate of adverse reactions | Immediately after follow-up check
  Rate of adverse reactions
Patient compliance | Immediately after follow-up check
  good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Derived] Kong Q, Mirza IA, Zhang X, Song X, Li X, Zhang Q, Xu L, Guo Y, Yu Y, Zuo X, Li Y, Li Y. Fourteen-Day Tegoprazan-Amoxicillin Dual Therapy as the First-Line Treatment of Helicobacter pylori Infection (SHARE2301): A Multicenter, Noninferiority, Randomized Clinical Trial. Helicobacter. 2024 May-Jun;29(3):e13098. doi: 10.1111/hel.13098. PMID 38853394